CLINICAL TRIAL: NCT00273637
Title: Pregnancy Related Cardiomyopathy Enrollment and Lessons in Web-Based Recruitment (PRiCELESS)
Brief Title: Registry and Survey of Women With Pregnancy Related Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Vincent's Medical Center (Unknown)
Organization: St Vincent's Hospital (Other)
Other Study IDs: STVincentH
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2005-10

CONDITIONS: Cardiomyopathy; Pregnancy-Associated Cardiomyopathy; Heart Failure
Keywords: heart failure; peripartum cardiomyopathy; pregnancy-associated cardiomyopathy; pregnancy complications; nonischemic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies; Peripartum Cardiomyopathy; Heart Failure; Pregnancy Complications

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The goal of this study is to better characterize peripartum cardiomyoapthy or pregnancy-related cardiomyopathy by enrolling as many PPCM survivors as possible using both direct and web-based methods of recritment. Patients will anser a questionnaire regarding the onset, progression, treatment and follow-up of their diagnosis as well as the psychosocial aspects of PPCM.

DETAILED DESCRIPTION:
The design of our study will utilize web-based recruitment methods with internet-based support groups for PPCM e.g. www.AMothersHeart.org (www.amothersheart.org/index.html). The directors of these websites will facilitate contact between our research staff and the several hundred members of these web sites.

An introductory letter will be posted on the website introducing the cardiovascular research team and describing the purpose, basic methods, and goals of our study. Website members who desire to participate can respond to a dedicated e-mail address we have set up and provide contact information so that we may get informed consent via telephone or mailed written consent. A telephone number will also be provided for participants so that they may call with questions regarding the study. Patients will then receive a questionnaire addressing our study goals. Questions will focus on obtaining family and social history, characterizing presenting symptoms, initial management, and clinical course following delivery of the fetus including extent of cardiovascular follow-up, date of echocardiograms performed, medications, and psychosocial support, if provided.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if diagnosed with PPCM after January 1, 1994. Patients must be above the age of 18 years old with no prior cardiac history and no history of chronic drug or alcohol abuse. Diagnosis of PPCM must have been made prior after the 28th week of gestation and up to 6 months postpartum. Patients must have echocardiographic data confirming left ventricular systolic dysfunction by either depressed shortening fraction or depressed ejection fraction.

Exclusion Criteria:

Patients with an identifiable etiology for their heart failure will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175
Dates: Start 2005-10; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Jordan G Safirstein, MD, Principal Investigator — Saint Vincent's Catholic MEdical Center; Cezar Staniloae, MD, FACC, Study Director — SVCMC
Locations (1):
- Saint Vincent's Catholic Medical Center, New York, New York, United States

REFERENCES:
- [Background] Ro A, Frishman WH. Peripartum cardiomyopathy. Cardiol Rev. 2006 Jan-Feb;14(1):35-42. doi: 10.1097/01.crd.0000174805.68081.f7. PMID 16371764
- [Background] Fett JD, Christie LG, Carraway RD, Murphy JG. Five-year prospective study of the incidence and prognosis of peripartum cardiomyopathy at a single institution. Mayo Clin Proc. 2005 Dec;80(12):1602-6. doi: 10.4065/80.12.1602. PMID 16342653